CLINICAL TRIAL: NCT00312481
Title: A Randomised, Single-Centre, Parallel-Group, Pilot Study to Assess the Efficacy, Safety and Patient Acceptability of a New 2-Litre Bowel Preparation Agent (MOVIPREP®) Compared With a Standard Bowel Preparation Agent (PICOLAX®)
Brief Title: MOVIPREP® Versus PICOLAX® Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Dr Mike Geraint, Norgine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NRL994-02-2004
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Colonoscopy
MeSH Terms: interventions — MoviPrep

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MOVIPREP
  Interventions: Drug: macrogol3350 NA sulphate NACL KCL ascorbic acid NA ascorbate
- 2 (Active Comparator): Picolax
  Interventions: Drug: NA picosulfate magnesium citrate

INTERVENTIONS:
Drug: macrogol3350 NA sulphate NACL KCL ascorbic acid NA ascorbate — Split dose, 1-litre solution in the evening prior to colonoscopy and second dose in the morning prior to colonoscopy
  Other Names: MOVIPREP
  Arms: 1
Drug: NA picosulfate magnesium citrate — 150 ml solution before 8am on day prior to colonoscopy and 150ml solution 6 to 8 hours later.
  Arms: 2

SUMMARY:
This will be a randomised, single-centre, single-blind, parallel-group, pilot study in patients undergoing colonoscopy.

The primary objective is to evaluate the efficacy of MOVIPREP® versus PICOLAX® for gut cleansing prior to colonoscopy.

The secondary objectives are to evaluate the safety, tolerability and acceptability of MOVIPREP versus PICOLAX for gut cleansing prior to colonoscopy.

DETAILED DESCRIPTION:
Gut cleansing will be performed using a split dose of MOVIPREP®, 1-litre solution (1x sachet A and 1x sachet B) in the evening prior to the day of colonoscopy and 1-litre solution (1x sachet A and 1x sachet B) in the morning of the colonoscopy, or PICOLAX®, 150 mL solution (1 sachet) before 8am on day prior to the day of colonoscopy, and 150 mL solution (1 sachet) 6 to 8 hours later.

The primary efficacy measure will be the degree of gut cleansing, as assessed by the physician performing the colonoscopy. A 5-grade scale will be used to assess each of the predefined colon areas, resulting in a final grading (A to D) of the overall quality of the bowel preparation treatment. Grades A and B will be considered as success, and Grades C and D as failure.

The secondary efficacy measures will be:

* is it necessary for the patient to return for a further colonoscopy due to insufficient clearance/cleansing of colon prior to the normal schedule for a repeat procedure?
* taste acceptability
* ease of taking, and ability to complete the bowel preparation treatment
* recommended diet compliance
* would the patient be prepared to repeat the bowel preparation treatment if necessary?
* well-being and effect on usual activities whilst taking the bowel preparation treatment
* overall impression of the bowel preparation treatment prior to colonoscopy
* symptoms experienced since taking their first study bowel preparation treatment and prior to their colonoscopy

Safety and tolerability will be assessed through the collection of adverse events, clinical laboratory tests, physical examination, weight and vital signs (blood pressure and pulse rate) data.

Number of patients:

It is intended to recruit approximately 70 patients in order to achieve at least 60 evaluable patients using a randomisation ratio of 1:1 MOVIPREP®: PICOLAX®.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent obtained prior to inclusion
* male or female, aged 18 to 80 years, inclusive, scheduled to undergo a complete colonoscopy
* willing, able and competent to complete the entire procedure and to comply with study instructions
* females of childbearing potential must employ an adequate method of contraception
* if an adequate method of contraception is not being used, the patient will be post hysterectomy, post bilateral oophorectomy, post menopause or have any other condition which precludes pregnancy
* females of childbearing potential must undergo a pregnancy test

Exclusion Criteria:

* ileus
* gastro-intestinal obstruction or perforation
* toxic megacolon, toxic colitis
* congestive heart failure (New York Heart Association [NYHA] III + IV)
* acute life-threatening cardiovascular disease
* acute surgical abdominal conditions
* untreated or uncontrolled arterial hypertension
* known clinically significant reduced renal function with creatinine > 170 µmol/L
* known clinically significant reduced liver function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2005-07; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Overall quality of the bowel preparation treatment, based on the degree of gut cleansing of each section of the colon. | 8 days

SECONDARY OUTCOMES:
is it necessary for the patient to return for a further colonoscopy due to insufficient clearance/cleansing of colon prior to the normal schedule for a repeat procedure? | within 3 months
taste acceptability | 8 days
ease of taking, and ability to complete, the bowel preparation treatment | 8 days
recommended diet compliance | 8 days
would the patient be prepared to repeat the bowel preparation treatment if necessary? | 8 days
well-being and effect on usual activities whilst taking the bowel preparation treatment | 8 days
overall impression of the bowel preparation treatment prior to colonoscopy | 8 days
symptoms experienced since taking their first study bowel preparation treatment and prior to their colonoscopy | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Mike Geraint, MD, Study Director — Norgine
Locations (1):
- John Radcliffe Hospital, Department of Gastroenterology, Endoscopy Unit, Headley Way, Headington, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Hookey LC, Depew WT, Vanner SJ. A prospective randomized trial comparing low-dose oral sodium phosphate plus stimulant laxatives with large volume polyethylene glycol solution for colon cleansing. Am J Gastroenterol. 2004 Nov;99(11):2217-22. doi: 10.1111/j.1572-0241.2004.40482.x. PMID 15555005
- [Derived] Worthington J, Thyssen M, Chapman G, Chapman R, Geraint M. A randomised controlled trial of a new 2 litre polyethylene glycol solution versus sodium picosulphate + magnesium citrate solution for bowel cleansing prior to colonoscopy. Curr Med Res Opin. 2008 Feb;24(2):481-8. doi: 10.1185/030079908x260844. PMID 18179734